CLINICAL TRIAL: NCT03989440
Title: A Multicenter, Two Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AXER-204 in Subjects With Chronic Spinal Cord Injury
Brief Title: AXER-204 in Participants With Chronic Spinal Cord Injury
Acronym: RESET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ReNetX Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RNX-AX204-101
Record Dates: First submitted 2019-06-11; First posted 2019-06-18 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Chronic Spinal Cord Injury
Keywords: myelin-associated inhibitor; Nogo-A; MAG; OMgp; Nogo Receptor

STUDY DESIGN:
Intervention Model Description: Part 1 is open-label single-ascending dose. Part 2 is double-blind, placebo-controlled, repeat dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 - None; Part 2 - Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXER-204 (Experimental): Part 1 - Single ascending doses; Part 2 - Repeated dose
  Interventions: Drug: AXER-204
- Placebo (Placebo Comparator): Part 2 only - Repeated dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXER-204 — human NoGo Trap fusion protein
  Other Names: human NoGo Trap; human Nogo Receptor decoy
  Arms: AXER-204
Drug: Placebo — Phosphate buffered saline formulation
  Arms: Placebo

SUMMARY:
This two-part trial will assess the safety, tolerability, pharmacokinetics, and efficacy of AXER-204 administered by lumbar puncture and slow bolus infusion. Part 1 will evaluate the safety, tolerability, and pharmacokinetics of single ascending doses of AXER-204. Part 2 will evaluate the safety, tolerability, pharmacokinetics, and efficacy of repeated doses AXER-204 in comparison to placebo.

DETAILED DESCRIPTION:
AXER-204 is a human fusion protein that acts as a soluble decoy/trap for the myelin-associated inhibitors of axonal growth known as Nogo-A, MAG, and OMgp. AXER-204 and a surrogate protein used in early preclinical studies have been found to promote axon growth and recovery of function in animal models of spinal cord injury.

Part 1 of the trial is a multicenter, open-label, single ascending dose study in participants with chronic cervical spinal cord injury. Four cohorts of 6 participants each are planned, with participants within each cohort expected to receive the same dose of AXER-204.

Part 2 is a multicenter, randomized, double-blind, placebo-controlled, repeat dose study in chronic cervical spinal cord injury participants. Approximately 32 participants will be randomized (ratio 1:1) to receive repeated doses of AXER-204 or placebo (a phosphate buffered saline formulation). The dose level and dose frequency will be dependent upon outcomes from Part 1.

ELIGIBILITY:
Key Inclusion Criteria:

1. Traumatic spinal cord injury that occurred ≥ 1 year ago
2. Cervical spinal cord injury with serious neurologic deficit as evidenced by 1) bilateral ISNCSCI UEMS between 4 and 36 points inclusive, and 2) bilateral GRASSP Prehension Ability score between 4 and 17 points inclusive
3. Confirmation by MRI of the following:

   1. Chronic SCI (persistent spinal cord lesion)
   2. For AIS grade of A without sensory or motor zone of partial preservation extending at least two levels caudal to the level of injury, no apparent transection of the cord
   3. CSF space spanning the lesion

Key Exclusion Criteria:

1. Penetrating injury to the cord or spinal cord trauma caused by ballistic injury including gunshot that did not penetrate the spinal cord
2. History of stroke, cerebrovascular injury, or elevated intracranial pressure
3. Contraindications for lumbar puncture
4. Requiring mechanical ventilatory assistance of any type
5. Body mass index (BMI) ≥ 35 kg/m2 or body weight <50 kg
6. History of life threatening allergic or immune-mediated reaction to vaccines, or biologic drugs, at any time or any life threatening allergic or immune-mediated reaction within the past 12 months
7. Subjects fitted with an implanted pump or port for delivery of therapeutics to the CSF
8. Uncontrolled medical condition including but not limited to cardiovascular disease, sleep apnea, obstructive lung disease, severe neuropathic or severe chronic pain, severe autonomic dysreflexia
9. Participation in any other investigational drug or device trial within 30 days or within 5 half-lives of the investigational drug or any past participation in a SCI cellular therapy trial.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Maynard, PhD, Study Director — ReNetX Bio
Locations (6):
- United States (6):
  - Keck Medicine of USC, Los Angeles, California
  - Shepherd Center, Atlanta, Georgia
  - Shirley Ryan AbilityLab / Northwestern, Chicago, Illinois
  - Spaulding Rehabilitation, Boston, Massachusetts
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Maynard G, Kannan R, Liu J, Wang W, Lam TKT, Wang X, Adamson C, Hackett C, Schwab JM, Liu C, Leslie DP, Chen D, Marino R, Zafonte R, Flanders A, Block G, Smith E, Strittmatter SM. Soluble Nogo-Receptor-Fc decoy (AXER-204) in patients with chronic cervical spinal cord injury in the USA: a first-in-human and randomised clinical trial. Lancet Neurol. 2023 Aug;22(8):672-684. doi: 10.1016/S1474-4422(23)00215-6. PMID 37479373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1: 25 participants were enrolled. One patient was withdrawn from the study prior to dosing and is not included in the Safety Population used for data analyses. Part 2: 27 participants were enrolled.
Groups:
- Part 1 - AXER-204 - 3 mg; Part 1 - AXER-204 - 30 mg; Part 1 - AXER-204 - 90 mg; Part 1 - AXER-204 - 200 mg: Part 1 Open-label single ascending dose. Participants received a single dose of AXER-204. AXER-204: human NoGo Trap fusion protein
- Part 2 - AXER-204 - 200 mg: Part 2 Double-blind, placebo-controlled repeat dose. Participants received up to 6 doses given approximately every 21 days. AXER-204: human NoGo Trap fusion protein
- Part 2 - Placebo: Part 2 Double-blind, placebo-controlled repeat dose. Participants received up to 6 doses given approximately every 21 days. Placebo: Phosphate buffered saline formulation
Period: Overall Study
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Started | 6 | 6 | 6 | 7 | 14 | 13
Completed | 6 | 6 | 5 | 6 | 14 | 13
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — COVID-19 travel restrictions | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unsuccessful lumbar puncture | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 13 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 00 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 14 | 12 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (9.1) | 44.8 (11.5) | 37.3 (16) | 41.2 (16.2) | 41.1 (13.8) | 34.5 (13.2) | 38.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 1 | 3 | 10
  Male | 5 | 6 | 5 | 2 | 13 | 10 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 1 | 2 | 7
  White | 3 | 5 | 5 | 5 | 12 | 11 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 14 | 13 | 51
International Standards for the Neurological Classification of Spinal Cord Injury, Bilateral Upper E [Mean (Standard Deviation); unit: units on a scale] — The ISNCSCI bilateral Upper Extremity Motor Score (UEMS) is determined by examining the muscle function within each of the 5 myotomes encompassing arm and hand function on each side of the body. A score ranging from 0 to 5 can be given to each myotome tested resulting in a maximum score of 50. Higher values indicate greater strength.
  units on a scale | 24.2 (6.6) | 26.7 (6.3) | 28.0 (5.5) | 28.7 (4.8) | 26.6 (5.4) | 23.9 (5.6) | 26.1 (5.6)
Graded Redefined Assessment of Strength, Sensibility, and Prehension; Bilateral Prehension Performan [Mean (Standard Deviation); unit: units on a scale] — The GRASSP Bilateral Prehension Performance Score is determined based on performance of four tasks with each hand with scores ranging from 0 to 5 for each task resulting in a maximum score of 40. Higher scores indicate better function.
  units on a scale | 16.5 (5.8) | 21.0 (7.6) | 18.0 (6.3) | 16.3 (6.7) | 16.4 (3.8) | 18.5 (4.5) | 17.7 (5.4)
Spinal Cord Independence Measure, Version III; Self-care [Mean (Standard Deviation); unit: units on a scale] — The SCIM III questionnaire self-care score assesses activities of daily living including feeding, bathing, dressing, and grooming. The self-care score ranges 0-20 with higher scores correspond to better ability to carry out these self-care activities.
  units on a scale | 9.8 (5.0) | 8.5 (4.7) | 11.5 (2.8) | 10.3 (3.6) | 10.4 (5.7) | 11 (3.6) | 10.4 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, or is a medically important event.
Time Frame: Up to Day 29 for Part 1 and Day 253 for Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 13
Participants | 5 | 4 | 5 | 6 | 14 | 10

2. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of AXER-204 in Serum
Time Frame: Part 1: pre-dose and 1 h, 6 h, 12 h, and 24 h post-dose, Day 4, 8, 15, and 29, Part 2: pre-dose and 4 h post-dose on days 1, 21, 42, 63, and 104; and on Study Days 169 and 253.
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
h*ng/mL | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | 3670 (1520) | 20900 (7540) | NA (NA) — Could not be calculated due to the limited sampling interval |

3. Primary Outcome: Cmax in Serum
Time Frame: as for outcome 2
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
ng/mL | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit determination | 277 (79.1) | 641 (173) | NA (NA) — Could not be determined due to the limited sampling interval |

4. Primary Outcome: Tmax in Serum
Time Frame: as for outcome 2
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
hours | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit determination | 16.8 (6.5) | 12.8 (5.06) | NA (NA) — Could not be determined due to the limited sampling interval |

5. Primary Outcome: t1/2 in Serum
Time Frame: as for outcome 2
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
hours | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | 53.9 (24.8) | NA (NA) — Could not be calculated due to the limited sampling interval |

6. Primary Outcome: Clearance From Serum
Time Frame: Day 1 pre-dose up to Day 29 in Part 1, Pre-dose up to Day 253 in Part 2
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
L/h | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | 4.84 (1.41) | NA (NA) — Could not be calculated due to the limited sampling interval |

7. Primary Outcome: Volume of Distribution
Description: Volume of distribution calculated from serum exposure data
Time Frame: as for outcome 2
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
L | NA (NA) — All values below limit of quantification | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | 344 (70.1) | NA (NA) — Could not be calculated due to the limited sampling interval |

8. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time of the Last Measurable Concentration (AUClast) of AXER-204 in CSF
Time Frame: Part 1: pre-dose, post-dose at 24 h, 72 h, Days 8 and 29, Part 2: pre-dose on Days 1, 21, 42, 63, and 104, and on Day 253.
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
h*ng/mL | 57200 (61500) | 5810000 (12300000) | 12500000 (18000000) | 10000000 (6260000) | NA (NA) — Could not be calculated due to the limited sampling interval |

9. Primary Outcome: Cmax of AXER-204 in CSF
Time Frame: as for outcome 8
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
ng/mL | 3340 (2890) | 87900 (128000) | 280000 (221000) | 412000 (129000) | NA (NA) — Could not be determined due to the limited sampling interval |

10. Primary Outcome: Tmax of AXER-204 in CSF
Time Frame: as for outcome 8
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
h | 24.2 (0.91) | 23.9 (0.89) | 23.2 (0.49) | 22.9 (0.93) | NA (NA) — Could not be determined due to the limited sampling interval |

11. Primary Outcome: t1/2 of AXER-204 in CSF
Time Frame: as for outcome 8
Population: In Part 2, only pharmacokinetic samples from participants receiving AXER-204 were analyzed (n=14).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 14 | 0
h | NA (NA) — Quantifiable concentrations were present in too few of the samples to permit calculation | 23.1 (32.2) | 13.5 (10.8) | 12.5 (7.08) | NA (NA) — Could not be calculated due to the limited sampling interval |

12. Secondary Outcome: Change in International Standards for Neurological Classification of SCI (ISNCSCI) Bilateral Upper Extremity Motor Score (UEMS)
Description: The ISNCSCI bilateral Upper Extremity Motor Score (UEMS) is determined by examining the muscle function within each of the 5 myotomes encompassing arm and hand function on each side of the body. A score ranging from 0 to 5 can be given to each myotome tested resulting in a maximum score of 50. Higher values indicate greater strength.
Time Frame: Baseline to Day 169
Population: This was pre-specified to be an exploratory outcome in Part 1, and therefore data will not be reported
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 14 | 13
score on a scale | 2.05 [0.59 to 3.52] | 1.52 [0.021 to 3.01]
Statistical Analysis 1: Comparison: Part 2 - AXER-204 - 200 mg vs Part 2 - Placebo; Test type: Superiority; p = 0.59, Mixed Models Analysis; LS Mean Difference = 0.54, 95% CI 2-sided [-1.48 to 2.55]

13. Secondary Outcome: Change in Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) Bilateral Prehension Performance Score
Description: The GRASSP Bilateral Prehension Performance Score is determined based on performance of four tasks with each hand with scores ranging from 0 to 5 for each task resulting in a maximum score of 40. Higher scores indicate better function.
Time Frame: Baseline to Day 169
Population: This was pre-specified to be an exploratory outcome in Part 1, and therefore data will not be reported
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 14 | 13
score on a scale | 0.42 [-1.07 to 1.91] | 1.97 [0.41 to 3.54]
Statistical Analysis 1: Comparison: Part 2 - AXER-204 - 200 mg vs Part 2 - Placebo; Test type: Superiority; p = 0.13, Mixed Models Analysis; LS Mean Difference = -1.56, 95% CI 2-sided [-3.62 to 0.50]

14. Secondary Outcome: Change in Version III of the Spinal Cord Independence Measure (SCIM III) Self-care
Description: The SCIM III questionnaire self-care score assesses activities of daily living including feeding, bathing, dressing, and grooming. The self-care score ranges 0-20 with higher scores correspond to better ability to carry out these self-care activities.
Time Frame: Baseline to Day 169
Population: This was pre-specified to be an exploratory outcome in Part 1, and therefore data will not be reported
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 14 | 13
score on a scale | -0.25 [-1.50 to 1.00] | 0.91 [-0.38 to 2.20]
Statistical Analysis 1: Comparison: Part 2 - AXER-204 - 200 mg vs Part 2 - Placebo; Test type: Superiority; p = 0.16, Mixed Models Analysis; LS Mean Difference = -1.16, 95% CI 2-sided [-2.81 to 0.50]

15. Secondary Outcome: Patient Global Impression of Change (PGIC) Responder Rate
Description: The PGIC instrument captures the patient's overall evaluation of response to treatment. Specifically, the PGIC asks: "Since beginning this clinical trial, how would you describe the overall change (if any) related to your chronic spinal cord injury?" The patient is asked to report the degree to which they have changed since entering the treatment period using a 7-point Likert scale (1='Much worse', 2='Worse', 3='A little worse', 4='No change', 5='A little better', 6='Better', 7='Much better') and "If better or worse, what has changed?". Patients that have evaluation results including "Much better", "Better", or "A little better" are considered Responders.
Time Frame: Day 169
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 14 | 13
Participants | NA — Not evaluated in Part 1 | NA — Not evaluated in Part 1 | NA — Not evaluated in Part 1 | NA — Not evaluated in Part 1 | 3 | 4
Statistical Analysis 1: Comparison: Part 2 - AXER-204 - 200 mg vs Part 2 - Placebo; Test type: Superiority; p = 0.68, Fisher Exact; % Difference in responder rate = -9.3, 95% CI 2-sided [-43.3 to 25.4]

ADVERSE EVENTS:
Time Frame: Part 1: up to Day 29, Part 2: up to Day 253
Arm/Group | Part 1 - AXER-204 - 3 mg | Part 1 - AXER-204 - 30 mg | Part 1 - AXER-204 - 90 mg | Part 1 - AXER-204 - 200 mg | Part 2 - AXER-204 - 200 mg | Part 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 4/14 | 2/13
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 5/6 | 6/6 | 14/14 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - AXER-204 - 3 mg (N=6) | Part 1 - AXER-204 - 30 mg (N=6) | Part 1 - AXER-204 - 90 mg (N=6) | Part 1 - AXER-204 - 200 mg (N=6) | Part 2 - AXER-204 - 200 mg (N=14) | Part 2 - Placebo (N=13)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - AXER-204 - 3 mg (N=6) | Part 1 - AXER-204 - 30 mg (N=6) | Part 1 - AXER-204 - 90 mg (N=6) | Part 1 - AXER-204 - 200 mg (N=6) | Part 2 - AXER-204 - 200 mg (N=14) | Part 2 - Placebo (N=13)
Headache (Nervous system disorders) | 3 | 1 | 3 | 5 | 13 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 2 | 3 | 5
Pleocytosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 6 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0 | 1 | 4 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 6 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 3 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 3
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1
CSF protein increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
CSF white blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 2 | 1
Mental fatigue (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Labile hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are free to publish, present, or use institution specific study data and results arising out of their performance of the protocol. At least forty five (45) days prior to submission for publication, PIs must submit to sponsor for review and comment any proposed oral or written publication. The first publication of the results shall be a joint multi-center publication of the study results managed and coordinated by sponsor unless this is not completed within 18 months after completion date.

DOCUMENTS (3):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03989440/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03989440/SAP_001.pdf
  • Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03989440/ICF_002.pdf